CLINICAL TRIAL: NCT05225610
Title: Comparison of Valsalva Manoeuvre and Intravenous Dexmedetomidine on Attenuating Pain During Propofol Injection in Upper Gastrointestinal Endoscopy: A Prospective Randomized Controlled Study
Brief Title: Valsalva Manoeuvre and Intravenous Dexmedetomidine on Attenuating Pain During Propofol Injection in Upper GIT Endoscopy
Acronym: Valsalva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, AHMED ABDELAZIZ SHAMA, LECTURER OF ANESTHESIA AND SURGICAL ICU, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRC13412/02/9
Record Dates: First submitted 2022-02-01; First posted 2022-02-04 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Injection Site Irritation
Keywords: Propofol injection pain; Dexmedetomidine; Valsalva Maneuver
MeSH Terms: interventions — Valsalva Maneuver; Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VALSALVA Group (Experimental): 40 Patients will perform the Valsalva manoeuvre before starting propofol injection by blowing into rubber tubing connected to a sphygmomanometer and raising the mercury column to 30 mmHg for at least 20 seconds and 5 ml saline will be administered in 5 seconds.
  Interventions: Other: Valsalva Manoeuvre
- DEXMED Group (Experimental): 40 patients will receive the tube between the lips, however, the manoeuvre will not be performed in this group, patients will receive 0.5 µg/kg Dexmedetomidine diluted in 5 ml saline in 5 seconds as a sedating dose prior to injection of propofol.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- CONTROL Group (Placebo Comparator): 40 patients will receive the tube between the lips, however, the manoeuvre will not be performed in this group and only 5 ml saline will be administered over 5 seconds.
  Interventions: Drug: normal Saline

INTERVENTIONS:
Other: Valsalva Manoeuvre — Blowing into rubber tubing connected to a sphygmomanometer and raising the mercury column to 30 mmHg for at least 20 seconds
  Arms: VALSALVA Group
Drug: Dexmedetomidine Injection [Precedex] — The study drugs will be kept at room temperature, preservative-free and will be prepared by an independent anaesthetist into 5 ml of total volume with the addition of 0.9 % normal saline. Tourniquet will be left inflated for 1 minute. Dexmedetomidine mixture and saline will be injected over 5 seconds. After the injection of the drugs, the tourniquet will be released
  Other Names: Precedex
  Arms: DEXMED Group
Drug: normal Saline — 5 ml saline will be administered.
  Other Names: saline
  Arms: CONTROL Group

SUMMARY:
No previous study has cited the use of the Valsalva manoeuvre for the reduction of pain on propofol injection in comparison with dexmedetomidine injection. Therefore, investigators plan a study to evaluate the analgesic efficacy of the Valsalva manoeuvre in alleviating pain during propofol injection as compared to dexmedetomidine injection.

DETAILED DESCRIPTION:
Propofol is a commonly used anaesthetic for inducing general anaesthesia. Pain on propofol injection is distressing and is one of the limitations of its use. Propofol is a phenol compound, which irritates nerve endings on the venous endothelium to produce immediate pain, whereas delayed pain is mediated by the release of bradykinin. Bradykinin causes vasodilation and increases venous permeability, thereby facilitating contact of the aqueous phase of propofol with nerve endings. Delayed pain occurs 10-20 seconds after injection.

Various methods have been tried so far to reduce pain on propofol injection. A commonly used technique is lignocaine either as pre-treatment or mixed with propofol. Other methods include the use of butorphanol, ondansetron, metoclopramide, opioid, or thiopentone. Propofol injection into a large vein, pre-injection cooling, or warming of propofol have also been investigated.

The Valsalva manoeuvre is a physiological technique, used in the reduction of pain associated with several procedures. The Valsalva manoeuvre alleviates both the somatic and psychological aspects of painful procedures.

Dexmedetomidine is an alpha-2 adrenoceptor agonist that has analgesic and sedative properties, it has been evaluated for reducing the incidence and intensity of propofol-induced pain, but reported results are inconsistent.

in this study, investigators will study the effect of Valsalva manoeuvre as compared with dexmedetomidine injection in reducing the pain associated with propofol injection in upper gastrointestinal endoscopies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 30-60 years old.
2. American Society of Anesthesiologist physical status(ASA) Grade I and II.
3. Upper gastrointestinal Endoscopies.

Exclusion Criteria:

1. Patients with mental illness, restlessness.
2. Cardio-respiratory disease.
3. Chronic pain disorder.
4. Use of preoperative analgesic medication.
5. History of propofol allergy.
6. History of drug abuse.
7. Inability to perform the Valsalva manoeuvre. -

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-19 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 20 seconds after propofol injection.
  using a ruler as the visual analogue scale(VAS), The VAS score ranged from 0-10, with 0 indicating no pain and 10 indicating the worst imaginable pain. Patients will be instructed to mark a point on the VAS ruler that represented the intensity of pain. The pain score was determined by measuring the distance in mm between 0 (no pain) and the mark will be indicated by the patient on the ruler.

SECONDARY OUTCOMES:
Withdrawal response score | 20 seconds after propofol injection
  withdrawal response will be assessed using standard questions including comfort during injection, verbal response, and behavioural signs (facial grimacing, arm withdrawal, or tears). the withdrawal response scoring will be graded on a 4-point scale: 0 = no pain, 1 = mild pain (pain reported only in response to questioning without any behavioural signs), 2 = moderate pain (pain reported in response to questioning and accompanied by behavioural signs or pain reported spontaneously without questioning), and 3 = severe pain (strong vocal response or response accompanied by facial grimacing, arm withdrawal, or tears).
Heart Rate(HR) beat / minute | 10 minutes
  the heart rate (HR) will be recorded before the Valsalva manoeuvre, at 1 minute, at 2 minutes after the manoeuvre, following propofol injection, and 5 minutes later on
Propofol injection site reaction | 24 hour
  the propofol injection site will be checked for signs of inflammation including oedema, pain, wheal, and flare
Non-invasive blood pressure(NIBP) mmHg | 10 minutes.
  Non-invasive blood pressure(NIBP) will be recorded before the Valsalva manoeuvre, at 1 minute, 2 minutes after the manoeuvre, following propofol injection, and 5 minutes later on.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED A SHAMA, MD, Principal Investigator — LECTURER OF ANESTHESIA AND SURGICAL ICU, TANTA UNIVERSITY, FACULTY OF MEDICINE
Locations (1):
- Sharurah Armed Forces Hospital, Sharurah, Najran Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No